CLINICAL TRIAL: NCT03178084
Title: The Effects of Maraviroc Versus Efavirenz in Combination With Zidovudine/Abacavir on the CD4/CD8 Ratio in Treatment-naïve HIV-infected Individuals
Brief Title: Effects of Maraviroc vs. Efavirenz on CD4/CD8 Ratio
Acronym: MeritRate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MeritRate
Record Dates: First submitted 2017-04-07; First posted 2017-06-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2017-06

CONDITIONS: HIV/AIDS
Keywords: HIV; CD4/CD8 ratio; immune recovery; maraviroc; efavirenz
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Maraviroc; Zidovudine; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Maraviroc (UK-427,857) QD + Zidovudine/Lamivudine BID (Experimental): Maraviroc (UK-427,857) 300 mg once daily added to Zidovudine/Lamivudine (300 mg/150 mg twice daily).
  Following a review of the interim analysis data, the DSMB recommended to terminate the UK-427,857 300 mg QD arm based on pre-specified protocol non-inferiority criteria not being met for the QD arm versus efavirenz
  Interventions: Drug: Maraviroc (UK-427,857) QD + Zidovudine/Lamivudine BID
- Efavirenz QD + Zidovudine/Lamivudine BID (Active Comparator): Efavirenz (600 mg once daily) added to Zidovudine/Lamivudine (300 mg/150 mg twice daily
  Interventions: Drug: Efavirenz QD + Zidovudine/Lamivudine BID
- Maraviroc (UK-427,857) BID + Zidovudine/Lamivudine BID (Experimental): Maraviroc (UK-427,857) 300 mg twice daily added to Zidovudine/Lamivudine (300 mg/150 mg twice daily)
  Interventions: Drug: Maraviroc (UK-427,857) BID + Zidovudine/Lamivudine QD

INTERVENTIONS:
Drug: Maraviroc (UK-427,857) QD + Zidovudine/Lamivudine BID — maraviroc (UK-427,857) 300 mg once daily added to zidovudine/lamivudine (300 mg/150 mg twice daily
  Arms: Maraviroc (UK-427,857) QD + Zidovudine/Lamivudine BID
Drug: Efavirenz QD + Zidovudine/Lamivudine BID — efavirenz (600 mg once daily) added to zidovudine/lamivudine (300 mg/150 mg twice daily)
  Arms: Efavirenz QD + Zidovudine/Lamivudine BID
Drug: Maraviroc (UK-427,857) BID + Zidovudine/Lamivudine QD — maraviroc (UK-427,857) 300 mg twice daily added to zidovudine/lamivudine (300 mg/150 mg twice daily
  Arms: Maraviroc (UK-427,857) BID + Zidovudine/Lamivudine BID

SUMMARY:
A low CD4/CD8 ratio is considered a surrogate marker of immunosenescence and is an independent predictor of non-AIDS-related morbidity and mortality. Given the strong clinical implications the impact of different regimens on the CD4/CD8 ratio recovery needs to be analyzed. The MERIT study is a completed a randomized, double-blind, multicenter phase IIb/III study with an open-label extension phase (240-week follow-up) to assess the efficacy of zidovudine/lamivudine in combination with maraviroc (MVC) or efavirenz (EFV) in treatment-naïve patients. Anonymised patient level data of the MERIT trial to compare the trajectories of the CD4/CD8 ratio of participants treated with maraviroc vs. efavirenz will be used.

DETAILED DESCRIPTION:
The Merit study was a randomized, double-blind, active-comparator multicenter, phase IIb/III study, treatment- naive patients (aged at least 16 years) with R5 HIV-1, and with plasma viral load (HIV-1 RNA) above 2000 copies/ml, who received MVC 300mg q.d., MVC 300mg b.i.d., or EFV 600mg q.d., each in combination with ZDV/3TC 300 mg/150mg b.i.d. Key exclusion criteria included prior treatment with EFV, ZDV, 3TC, or any antiretroviral for more than 14 days at any time, and evidence of resistance to EFV, ZDV, or 3TC, as indicated by the presence of at least one nucleoside-associated mutations conferring resistance to ZDV, or phenotypic resistance to ZDV, at least one mutation conferring resistance to 3TC or phenotypic resistance to 3TC, or at least one mutation responsible for EFV resistance or phenotypic resistance to EFV.

Following a planned analysis at week 16, the MVC q.d. arm was discontinued for not meeting prespecified efficacy criteria, and the study continued with two treatment arms. The sponsor was unblinded at the 48-week analysis time point, but the investigators and patients remained blinded until the 96-week analysis. The study was then fully unblinded following the last patient's 96-week visit, and patients were enrolled in a nominal 3-year open-label phase. Efficacy and safety data from the 240-week (nominal 5-year) study duration have been recently published (Cooper D. et al, AIDS 2014).

The longitudinal data of the Merit study (240-week follow-up) will be analysed. The current long-term follow-up of the MERIT study, the extensive registry of both AIDS and non-AIDS clinical events and the randomization to a therapeutic intervention including maraviroc, will allow to evaluate the effects of maraviroc vs. efavirenz on the CD4/CD8 ratio trajectories.

All randomized subjects included in MERIT will be included in this exploratory post hoc analysis. For the principal objective, longitudinal changes in CD4 and CD8 counts and in the CD4/CD8 ratio will be assessed using generalized estimating equations. Interaction terms will be created to assess whether these changes over time differed significantly between treatment arms. Kaplan-Meier methods will be used to calculate the rates of CD4/CD8 normalization at 0.4 and 1 cut-offs and cumulative probabilities. Cox proportional hazard models will be used to compare probabilities of CD4/CD8 normalization by treatment arm.

ELIGIBILITY:
All patients analysed in the Merit trial (Cooper, JAIDS 2010)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 721 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2016-11-05 (Actual); Study Completion 2017-03-07 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in CD4/CD8 ratio | From baseline to week 120

SECONDARY OUTCOMES:
Change From Baseline in CD8+ T cells | From baseline to week 120
Change From Baseline in CD4/CD8 ratio | From baseline to week 120

IPD SHARING:
Plan to Share IPD: No